CLINICAL TRIAL: NCT00002481
Title: Phase II Study of High-Dose Cytarabine, Cisplatin, and Dexamethasone Followed By Cyclophosphamide, Etoposide, Total Body Irradiation, and Autologous Bone Marrow Rescue in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy and Radiation Therapy Plus Bone Marrow Transplantation in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Luke's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077128; STLMC-ABMR-9001; NCI-V91-0112
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2001-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cisplatin; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Procedure: autologous bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Bone marrow transplantation may allow doctors to give higher doses of radiation therapy and chemotherapy and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose etoposide and cyclophosphamide plus total-body irradiation followed by bone marrow transplantation in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and activity of cyclophosphamide, etoposide, total body irradiation, and autologous bone marrow transplantation in patients with relapsed or refractory non-Hodgkin's lymphoma. II. Determine the feasibility of pretransplantation cytoreduction with a regimen of high-dose cytarabine, cisplatin, and dexamethasone in this patient population. III. Determine the feasibility of posttransplantation radiotherapy given to sites of residual disease (involved-field "boost" irradiation) in this patient population.

OUTLINE: Patients are stratified by disease status (refractory vs relapsed). Autologous bone marrow is harvested before cytoreduction or involved field radiotherapy (IFRT). Patients with marrow involvement who achieve marrow complete response after cytoreduction undergo harvest of bone marrow before IFRT. Patients receive cytoreduction comprising high-dose cytarabine IV over 1 hour every 12 hours, cisplatin IV over 10 hours, and dexamethasone three times daily on days 1 and 2. At 3 weeks, a second course is administered if tumor reduction is at least 25% and in the absence of unacceptable toxicity. Patients with involved sites 2 cm or greater in diameter at evaluation and previously unirradiated active disease sites, at least 90% of which can be treated with IFRT, undergo IFRT 5 days a week for 2 weeks beginning after cytoreduction and 3-5 weeks after harvest of bone marrow. Within 10 days after completion of IFRT, patients receive etoposide IV over 26 hours beginning on day -7, cyclophosphamide IV over 2 hours on days -6 to -4, and total body irradiation twice daily on days -3 and -2 and once on day -1. Bone marrow is reinfused on day 0. Eligible patients with residual disease at 3 months after transplantation undergo involved field "boost" irradiation to sites of residual disease.

PROJECTED ACCRUAL: Approximately 50 patients (25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven or unequivocal radiologic evidence of non-Hodgkin's lymphoma that has relapsed or is refractory after first-line chemotherapy Unequivocal radiologic evidence of relapse defined as the presence of enlarged (at least 2 cm diameter) lymph nodes by CT scan or lymphangiogram Biopsy of accessible lymph nodes to confirm relapse encouraged Low-, intermediate-, or high-grade disease Normal bilateral bone marrow biopsy at time of bone marrow collection required (cellularity at least 20% and no histologic evidence of tumor) History of marrow involvement allowed if present marrow is histologically normal No disease progression in a previously irradiated site A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: CALGB 0-2 Karnofsky 70-100% Life expectancy: More than 2 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 3 times normal SGOT and SGPT less than 3 times normal Alkaline phosphatase less than 3 times normal Hepatitis B surface antigen negative Renal: Creatinine normal Creatinine clearance at least 60 mL/min Cardiovascular: Cardiac ejection fraction normal by MUGA scan No uncontrolled or severe cardiovascular disease, including the following: Myocardial infarction within the past 6 months Congestive heart failure Symptomatic angina (despite optimal medical management) Life-threatening arrhythmia or hypertension Pulmonary: Pulmonary function tests (DLCO and spirometry) greater than 60% predicted Other: HIV negative No serious organ dysfunction (unless caused by lymphoma) No active bacterial, viral, or fungal infection No active peptic ulcer disease No uncontrolled diabetes mellitus No other malignancy except curatively treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer No other serious medical or psychiatric illness that would preclude study Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Prior nitrosourea allowed if cumulative dose no more than 600 mg/m2 Prior bleomycin allowed if cumulative dose no more than 300 units/m2 Prior doxorubicin allowed if cumulative dose no more than 450 mg/m2 No prior high-dose etoposide (more than 1,800 mg/m2) No prior high-dose cyclophosphamide (more than 100 mg/kg) No chemotherapy within 4 weeks (no melphalan, nitrosourea, or mitomycin within 6 weeks) prior to bone marrow collection No prior salvage therapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to liver or lung Prior other radiotherapy allowed if doses do not exceed the following limits: 1,400 cGy to the mediastinum 1,400 cGy to the whole abdomen 4,000 cGy to the CNS Surgery: Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-03

CONTACTS AND LOCATIONS:
Overall Officials: Robert F. Taylor, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- St. Luke's Medical Center, Milwaukee, Wisconsin, United States